CLINICAL TRIAL: NCT02066077
Title: The Efficacy And Cognitive Impairment Of Modified Electroconvulsive Therapy: A Randomized Clinical Trial And Its Standard Technology Promotion Research
Brief Title: The Efficacy And Cognitive Impairment Of Modified Electroconvulsive Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Tongji Hospital (Other); Huashan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SHDC12012109
Record Dates: First submitted 2014-02-13; First posted 2014-02-19 (Estimated); Last update posted 2018-04-23 (Actual); Status verified 2017-12

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Modified Electroconvulsive Therapy; Cognition; Memory
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Etomidate; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Bilateral temporal and propofol (Experimental): During the MECT treatment, electrodes are placed at bilateral temporal, with propofol 2mg/kg to Induce anesthesia.
  Interventions: Drug: Propofol; Device: Bilateral temporal MECT
- Bilateral temporal and etomidate (Experimental): During the MECT treatment, electrodes are placed at bilateral temporal, with etomidate 0.3mg/kg to Induce anesthesia.
  Interventions: Drug: Etomidate; Device: Bilateral temporal MECT
- The right temporal and propofol (Experimental): During the MECT treatment, electrodes are placed at the right temporal, with propofol 2mg/kg to Induce anesthesia.
  Interventions: Drug: Propofol; Device: The right temporal MECT
- The right temporal and etomidate (Experimental): During the MECT treatment, electrodes are placed at the right temporal, with etomidate 0.3mg/kg to Induce anesthesia.
  Interventions: Drug: Etomidate; Device: The right temporal MECT
- Bilateral frontal and propofol (Experimental): During the MECT treatment, electrodes are placed at bilateral frontal, with propofol 2mg/kg to Induce anesthesia.
  Interventions: Drug: Propofol; Device: Bilateral frontal MECT
- Bilateral frontal and etomidate (Experimental): During the MECT treatment, electrodes are placed at bilateral frontal, with etomidate 0.3mg/kg to Induce anesthesia.
  Interventions: Drug: Etomidate; Device: Bilateral frontal MECT
- Standard-therapy Group (Active Comparator): During the MECT treatment, electrodes are placed at bilateral temporal, with etomidate 0.3mg/kg to Induce anesthesia.
  Interventions: Drug: Etomidate; Device: Bilateral temporal MECT

INTERVENTIONS:
Drug: Etomidate
  Arms: Bilateral frontal and etomidate; Bilateral temporal and etomidate; Standard-therapy Group; The right temporal and etomidate
Drug: Propofol
  Arms: Bilateral frontal and propofol; Bilateral temporal and propofol; The right temporal and propofol
Device: Bilateral temporal MECT
  Arms: Bilateral temporal and etomidate; Bilateral temporal and propofol; Standard-therapy Group
Device: The right temporal MECT
  Arms: The right temporal and etomidate; The right temporal and propofol
Device: Bilateral frontal MECT
  Arms: Bilateral frontal and etomidate; Bilateral frontal and propofol

SUMMARY:
1. To determine the influencing factors of modified electroconvulsive therapy (MECT);
2. To determine the influencing factors and reversibility of the cognitive impairment caused by MECT;
3. To determine the duration of efficacy of MECT and its affecting factors.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years (when informed consent was got), male or female
* Meet International Classification of Diseases-10(ICD-10) diagnostic criteria for depression
* Scored 18 or above on the HAM-D Scale which included 17 items
* Clinical Global Impression(CGI)-severity score ≥ 4
* Provided written informed consent

Exclusion Criteria:

* Any depressive disorders not due to major depressive disorder
* Meet other diagnosis criteria in Diagnostic and Statistical Manual of Mental Disorders-IV-Test Revision(DSM-IV-TR) Axis I
* With a history of acute or chronic renal failure, liver cirrhosis or active hepatopathy
* With clinically significant abnormal results of laboratory test, which are considered to have impact on treatment efficacy and the safety of participants
* With a history of severe or unstable physical disease including nervous system disease and myocardial infarction
* Undergoing alcoholism or alcohol (or substance) abuse during 30 days or 6 months before the trial
* With no response to previous ECT treatment
* Received transcranial magnetic stimulation treatment in the last 6 months
* Allergic to propofol, etomidate and succinylcholine chloride
* During pregnancy or lactation
* With a history of stroke in the last month
* Enrolled in any other clinical trial 30 days prior to the baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2013-01-01; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Hamilton Depression Scale(HAMD) Scores | Change from Baseline in Hamilton Depression Scale scores at 7d, 14d, 21d, 28d, 35d, 42d and 180d after the last MECT session
Change in Wechsler Memory Scale (WMS) Scores as a Measure of Safety | Change from Baseline in Wechsler Memory Scale (WMS) Scores at 42d and 180d after the last MECT session

SECONDARY OUTCOMES:
Young Manic Rating Scale(MMSE) as a Measure for Evaluation of Mania State | 42d and 180d after the last MECT session
Resting-state/Task-state functional magnetic resonance imaging (fMRI) | Change form Baseline in Resting-state/Task-state fMRI Imging Results at 42d and 180d after the last MECT session
Change in Hamilton Anxiety Scale(HAMA) Scores | Change from Baseline in Hamilton Anxiety Scale Scores at 7d, 14d, 21d, 28d, 35d, 42d and 180d after the last MECT session
Change in Clinical Global Impression-severity of illness(CGI-SI) Scores as a Measure of Efficacy | Change from Baseline in CGI-SI Scores at 7d, 14d, 21d, 28d, 35d, 42d and 180d after the last MECT session
Change in Wisconsin Card Sorting Test(WCST) Scores as a Measure of Safety | Change from Baseline in Wisconsin Card Sorting Test(WCST) Scores at 42d and 180d after the last MECT session
Change in P300/P50 Event-Related Potentials(ERP) | Change from Baseline in P300/P50 Event-Related Potentials(ERP) at 42d and 180d after after the last MECT session

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, China